CLINICAL TRIAL: NCT06352632
Title: A Multi-faCtorial, mulTi-arm, Multi-staGe, Randomised, gLOBal Adaptive pLatform Trial for Stroke (ACT-GLOBAL)
Brief Title: ACT-GLOBAL Adaptive Platform Trial for Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Calgary (Other); Berry Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-GLOBAL_Master
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Adaptive Platform Trial; Blood Pressure; Tenecteplase; Ischaemic stroke; Intracerebral Haemorrhage
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebral Hemorrhage | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Adaptive Platform Trial evaluating multiple interventions in multiple states and domains
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IV thrombolysis domain (Experimental): This domain has a prospective, randomized, controlled, open-label, parallel group with blinded endpoint assessment (PROBE) design to optimize the use of intravenous Tenecteplase in participants with Acute Ischemic Stroke.
  Interventions: Drug: Standard-dose intravenous tenecteplase; Drug: Low-dose intravenous tenecteplase; Other: No intravenous tenecteplase
- Blood Pressure domain (Experimental): Third Enhanced Control of Hypertension and Thrombectomy Stroke Study (ENCHANTED3/MT) as a domain of ACT-GLOBAL to compare three BP lowering management strategies, that of conservative, moderate and intensive BP lowering in patients with Acute Ischaemic Stroke admitted to participating hospitals who has an elevated SBP after reperfusion therapy via Endovascular Thrombectomy, and reliably determine, which approach leads to improved functional outcome.
  Locally available and approved i.v. BP lowering agents can be used in this domain.
  Interventions: Other: Conservative Blood Pressure Control; Other: Moderate Blood Pressure Control; Other: Intensive Blood Pressure Control
- ACT-42 domain (Experimental): This domain has a Phase 2b, multicenter, prospective, randomized, open label, blinded-endpoint (PROBE) controlled single-dose adaptive design and aim to determine the efficacy and safety of NoNO-42 in participants with Acute Ischaemic Stroke selected for thrombolysis with or without Endovascular Thrombectomy.
  Interventions: Other: Placebo; Drug: NoNO-42
- INTERACT5 Domain (Experimental): This is a domain within the Intracerebral Haemorrhage State of the ACT-GLOBAL adaptive platform trial for stroke.
  The objective of this domain is to determine the efficacy of intravenous deferoxamine and low-dose oral colchicine, both individually and in combination, compared to standard of care alone, on improving functional outcome in patients with acute spontaneous supratentorial ICH.
  Interventions: Other: No deferoxamine mesylate and no colchicine; Drug: Deferoxamine mesylate only; Drug: Colchicine only; Drug: Both deferoxamine mesylate and colchicine

INTERVENTIONS:
Drug: Standard-dose intravenous tenecteplase — Standard-dose intravenous tenecteplase (0.25 mg/kg body weight); one-time IV bolus injection soon after randomisation
  Arms: IV thrombolysis domain
Drug: Low-dose intravenous tenecteplase — Low-dose intravenous tenecteplase (0.18 mg/kg body weight); one-time IV bolus injection soon after randomisation
  Arms: IV thrombolysis domain
Other: No intravenous tenecteplase — No intravenous tenecteplase only in subjects on direct oral anticoagulant (DOACs) or those planned for emergency endovascular thrombectomy (EVT)
  Arms: IV thrombolysis domain
Other: Conservative Blood Pressure Control — No or minimal Systolic Blood Pressure (SBP) control; SBP reduction by 5-10mmHg or a target of 175-180mmHg if very-high baseline SBP (≥180mmHg); the timing of administration of interventions is specified to be immediately after randomisation; the intervention target is to be achieved ideally at 1 hour after randomisation and maintained for 24 hours (or until hospital discharge or death if this should occur earlier)
  Arms: Blood Pressure domain
Other: Moderate Blood Pressure Control — SBP reduction by 10-20mmHg or a target of 160 ± 5, whichever is higher; no control if low-high baseline SBP (150-160mmHg); the timing of administration of interventions is specified to be immediately after randomisation; the intervention target is to be achieved ideally at 1 hour after randomisation and maintained for 24 hours (or until hospital discharge or death if this should occur earlier)
  Arms: Blood Pressure domain
Other: Intensive Blood Pressure Control — SBP reduction by 30-50mmHg or a target of 140±5 mmHg, whichever is higher after endovascular thrombectomy (EVT); the timing of administration of interventions is specified to be immediately after randomisation; the intervention target is to be achieved ideally at 1 hour after randomisation and maintained for 24 hours (or until hospital discharge or death if this should occur earlier)
  Arms: Blood Pressure domain
Other: Placebo — 100 mL of 0.9% normal saline, administered as a single IV infusion with a 20-minute dosing duration.
  Arms: ACT-42 domain
Drug: NoNO-42 — NoNO-42 at weight-based dosing - 2.6 mg/Kg, administered as a single IV infusion with a 20-minute dosing duration
  Arms: ACT-42 domain
Other: No deferoxamine mesylate and no colchicine — No deferoxamine mesylate and no colchicine
  Arms: INTERACT5 Domain
Drug: Deferoxamine mesylate only — Deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) and continued for 2 consecutive days
  Arms: INTERACT5 Domain
Drug: Colchicine only — 0.5mg of oral colchicine daily for 30 days
  Arms: INTERACT5 Domain
Drug: Both deferoxamine mesylate and colchicine — Deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) and continued for 2 consecutive days; plus 0.5mg of oral colchicine daily for 30 consecutive days
  Arms: INTERACT5 Domain

SUMMARY:
Stroke is causing 6.6 million deaths and is a major cause of disability worldwide in 2019. There remains an urgent need for interventions that improve outcomes which can be implemented with wide applicability for stroke. ACT-GLOBAL is a multi-factorial, multi-arm, multi-stage, randomised, global adaptive platform trial for stroke, aiming to identify the treatment/s associated with the highest chance of improving outcome in stroke patients. In ACT-GLOBAL multiple questions will be evaluated simultaneously and sequentially as data accrues and can evaluate interactions between different treatment options.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death, worldwide. It is also the second largest cause of disability-adjusted-life-years (DALYs) lost after ischaemic heart disease in developing countries, and third largest contributor to DALYs in developed countries (after ischaemic heart disease, low back and neck pain). In 2019, the absolute numbers of new strokes (12.2 million), stroke-related deaths (6.6 million), and people living with stroke (101.5 million) had increased globally from 1990 (70%, 43%, and 85% increases, respectively).

Steady progress has been made in establishing specific management strategies for patients affected by, or at high-risk of, stroke. Unfortunately, only a few acute treatments have been proven to be beneficial: thrombolysis, endovascular thrombectomy, hemicraniectomy, stroke unit care, and aspirin. There is a continued need for interventions that improve outcomes which can be implemented with wide applicability for stroke.

ACT-GLOBAL is an investigator-initiated, multi-factorial, multi-arm, multi-stage, randomised, global adaptive platform trial for stroke, aiming to find the treatment/s associated with the highest chance of improving outcome after stroke. In ACT-GLOBAL multiple questions will be evaluated simultaneously and sequentially as data accrues and can evaluate interactions between different treatment options.

Frequent adaptive analyses are conducted to assess whether a given intervention is superior, inferior, or equivalent either within a domain or for specific populations within the domain. Where it is anticipated that interactions between interventions in different domains may be likely, the statistical models will allow evaluation of such interactions. Each intervention within a domain with prospectively defined and mutually exclusive strata (sub-groups) of participants will be evaluated within the strata, while information from one stratum may be used (via 'borrowing') to contribute to the analysis of the effect of that intervention in other strata. Specific interventions or subgroups within overall populations may be dropped or cease to enrol, based on pre-specified rules.

The adaptive design allows new interventions or domains or both to be introduced. A Response Adaptive Randomisation algorithm may be used to preferentially randomize participants to interventions that appear to be performing better in domains where applicable.

Unlike traditional trial designs which explicitly prohibit co-enrollment of patients into different trials or multiple therapies, or use a factorial design, the adaptive platform design allows investigators to replicate the real-world environment to estimate possible synergy, competitive interference, or safety profiles of complex treatment protocols.

ELIGIBILITY:
Platform Inclusion Criteria:

1. Age ≥18 years
2. Clinical diagnosis of stroke

Platform Exclusion Criteria:

There are no platform level exclusion criteria

Each state and domain will specify additional inclusion and exclusion criteria in the respective Domain-Specific Registration. Patients who fulfill the overall platform criteria will be assessed for enrollment into each active domain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) scores | Platform level time frame: 90 days in Ischaemic Stroke State; 6 months in Intracerebral Haemorrhage State; Domain specific time frame may differ (details will be included in domain-specific registration)
  The mRS is a 7-outcome ordered categorical scale that assesses functional neurological status after stroke. It is not intended for use as a measure of historical functional status. It is well accepted as a standard outcome around the world in the stroke community, by patients and by regulatory authorities. The seven values and the clinical summary of the individual scores are summarized in the following:
  0 = No symptoms
  1. = No significant disability; able to carry out all usual activities
  2. = Slight disability; can look after own affairs, but unable to carry out all previous activities
  3. = Moderate disability; require some help
  4. = Moderately severe disability; unable to attend to own bodily needs without assistance
  5. = Severe disability; bedridden and requiring constant nursing care and attention
  6. = Dead

SECONDARY OUTCOMES:
Excellent functional neurological outcome | Platform level time frame: 90 days in Ischaemic Stroke State; 6 months in Intracerebral Haemorrhage State; Domain specific time frame may differ (details will be included in domain-specific registration)
  Excellent functional neurological outcome means modified Rankin scale (mRS) scores 0-1. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Independent functional neurological outcome | Platform level time frame: 90 days in Ischaemic Stroke State; 6 months in Intracerebral Haemorrhage State; Domain specific time frame may differ (details will be included in domain-specific registration)
  Independent functional neurological outcome means modified Rankin scale (mRS) scores 0-2. The minimum mRS is 0 (no symptoms) while the maximum mRS is 6 (death). The higher the mRS score is the worse outcome is.
Health Related Quality of Life | Platform level time frame: 90 days in Ischaemic Stroke State; 6 months in Intracerebral Haemorrhage State; Domain specific time frame may differ (details will be included in domain-specific registration)
  Health Related Quality of Life based on EuroQol 5 Dimension 5 Level (EQ-5D-5L).The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems.

OTHER OUTCOMES:
Mortality | Platform level time frame: 90 days in Ischaemic Stroke State; 6 months in Intracerebral Haemorrhage State; State and Domain specific time frame may differ (details will be included in domain-specific registration)
  Mortality status equals to death which will be collected at all visits during the trial period

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, MD, PhD, Principal Investigator — The George Institute; Bijoy Menon, MD, Principal Investigator — University of Calgary; Michael D Hill, MD, Principal Investigator — University of Calgary; Andrew Demchuk, MD, Principal Investigator — University of Calgary; Xiaoying Chen, PhD, Principal Investigator — The George Institute
Locations (2):
- The George Institute for Global Health, Sydney, New South Wales, Australia
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
After a domain is completed, the archived de-identified limited dataset of randomized participants will be transmitted to and stored in the ACT-GLOBAL Data Repository, for use by researchers. Data can be shared after publication of the main results unless specified otherwise in domain-specific registration.
Supporting Information: Study Protocol
Time Frame: Data can be shared after publication of the main results.
Access Criteria: Data can be shared after publication of the main results, based on approval of a submitted protocol to the Publication Committee and relevant ethics review. Data can be shared to bona fide researchers with experience in medical research, and with no conflict of interest that may potentially influence their interpretation of any analyses, and employed by a recognised academic institute, health service organisation, commercial research organisation of from the pharmaceutical industry. The data sharing will be only for analyses within the constraints of the consent under which the data were originally gathered consent.
  Data sharing with industry will be according to relevant contracts with appropriate approvals from all stake holders.

REFERENCES:
- See also: ACT-GLOBAL IV Thrombolysis Domain Registration Link — https://clinicaltrials.gov/study/NCT06320431
- See also: ACT-GLOBAL Blood Pressure Domain Registration Link — https://clinicaltrials.gov/study/NCT06352619
- See also: ACT-GLOBAL ACT-42 Domain Registration Link — http://clinicaltrials.gov/study/NCT06403267